CLINICAL TRIAL: NCT01465425
Title: Incidence and Significance of Extracolonic Findings on CT Colonography: Retrospective Analysis of "National CT Colonography Trial" Data
Brief Title: Extracolonic Findings on Computed Tomography (CT) Colonography
Acronym: ACRIN7151
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: American College of Radiology Imaging Network (Network)
Responsible Party: Sponsor
Other Study IDs: ACRIN 7151; A7151 (Other: ACRIN Foundation)
Record Dates: First submitted 2011-10-31; First posted 2011-11-04 (Estimated); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: Solitary Pulmonary Nodules; Multiple Pulmonary Nodules; Renal Neoplasms; Adrenal Gland Neoplasms; Aortic Aneurysm, Abdominal; Liver Neoplasms; Adnexal and Skin Appendage Neoplasms; Lymphadenopathy; Pancreatic Neoplasms
Keywords: extracolonic findings; ECFs; CT colonography; computed tomography colonography; National CT Colonography Trial; ACRIN 6664
MeSH Terms: conditions — Solitary Pulmonary Nodule; Multiple Pulmonary Nodules; Kidney Neoplasms; Adrenal Gland Neoplasms; Aortic Aneurysm, Abdominal; Liver Neoplasms; Neoplasms, Adnexal and Skin Appendage; Lymphadenopathy; Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- E3/E4 Case Group: The Case Group will target consenting 141 participants from the cases with indeterminate but potentially significant findings (E3/E4s) other than pulmonary nodules.
- Pulmonary Nodules Case Group: The Pulmonary Nodules Case Group will comprise 119 cases with E3/E4 ECFs characterized as pulmonary nodules.
- E1 Control Group: The E1 Control Group will be drawn from the 866 E1 ECF cases from ACRIN 6664 to create a cohort of 260 E1 ECF cases. The Control Group for comparison with the Case Group and the Pulmonary Nodules Case Group will be selected at the Biostatistics and Data Management Center (BDMC). The BDMC will match E1 141 controls to the 141 case-group participants with indeterminate but potentially significant findings (E3/E4s). The BDMC will also match 119 E1 controls to the 119 E3/E4 pulmonary nodules cases. Controls will be matched by site, age caliper (5 years), and sex where possible.

SUMMARY:
The ACRIN 7151 trial will use medical records abstraction data from participants with extracolonic findings (ECFs) reported from the ACRIN 6664 National CT Colonography Trial to: 1) measure incidence of diagnostic imaging, hospitalization, and interventional procedures associated with ECFs reported on computed tomography colonography (CTC), delineated by type of ECF; 2) determine potential predictors of follow-up diagnostic imaging, hospitalization, and interventional procedures, delineated by type of ECF; and 3) evaluate the clinical/pathologic diagnoses associated with indeterminate but potentially significant ECFs. These data can be used to incorporate ECFs into existing models on the cost-effectiveness of CTC in colorectal cancer screening and can potentially be used to develop guidelines for the reporting and management of ECFs.

DETAILED DESCRIPTION:
The original ACRIN 6664 National CT Colonography Trial included 15 participating sites and a total study data set of 2531 participants. The target study data set for the ACRIN 7151 trial is 520 participants, assigned to one of three cohorts: an E3/E4 Case Group (n = 141) excluding pulmonary nodules, an E3/E4 Pulmonary Nodules Case Group (n = 119), and an E1 Control Group (n = 260) (see Section 8.6). Medical records will be collected by the site from their institutions and from the primary care provider identified by the participant during the ACRIN 6664 trial. Initial record collection will comprise the six months following CTC for all cohorts. Additional medical record collection (from other primary care providers, specialists, and hospitals, and for extended time periods) may be necessary for primary endpoint determination. ECFs are categorized according to the original radiology read of the CTC during the ACRIN 6664 trial.

ELIGIBILITY:
No participant sub-populations will be excluded prior to selection (the E1 population will be matched to the Case Group populations).

Data from the 15 participating sites from the ACRIN 6664 trial provide a study data set of 2531 participants, broken down into a total target study data set of 520 participants. Participants will be distributed into one of three cohorts as follows:

* The Case Group will target consenting 141 participants from the cases with indeterminate but potentially significant findings (E3/E4s) other than pulmonary nodules.
* The Pulmonary Nodules Case Group will comprise 119 cases with E3/E4 ECFs characterized as pulmonary nodules.
* The E1 Control Group will be drawn from the 866 E1 ECF cases to create a cohort of 260 E1ECF cases. The Control Group for comparison with the Case Group and the Pulmonary Nodules Case Group will be selected at the Biostatistics and Data Management Center (BDMC). The BDMC will match E1 141 controls to the 141 case-group participants with indeterminate but potentially significant findings (E3/E4s). The BDMC will also match 119 E1 controls to the 119 E3/E4 pulmonary nodules cases. Controls will be matched by site, age caliper (5 years), and sex where possible. Where an appropriate match cannot be obtained, the matching criteria will be relaxed. If potential participants decline study consent, we will then best-match additional cases for the appropriate group to maintain target populations. Any additional cases beyond the initial 520 participants identified for medical record collection will be matched as feasible.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All participants originally enrolled in the ACRIN 6664 National CT Colonography Trial are eligible for the ACRIN 7151 trial. The target study data set for the ACRIN 7151 trial is 520 participants, assigned to one of three cohorts: an E3/E4 Case Group (n = 141) excluding pulmonary nodules, an E3/E4 Pulmonary Nodules Case Group (n = 119), and an E1 Control Group (n = 260).
Sampling Method: Non-Probability Sample
Enrollment: 520 (Estimated)
Dates: Start 2011-09; Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Rates of Follow Up Imaging, Hospitalization, Intervention | 6 Months, 15 Months
  Estimate the rates of follow-up diagnostic imaging, hospitalization, and interventional procedures commonly associated with ECFs within six months of receiving CTC for all three cohorts (E3/E4, pulmonary nodules, and E1). Compare the rates of medical utilization among participants with indeterminate but potentially significant ECFs (E3/E4s) and participants with pulmonary nodules, to participants with no ECFs (E1s).

SECONDARY OUTCOMES:
Characterize Outcomes | 6 Months
  Categorize the outcome of potentially clinically significant findings detected by CTC into resolved and unresolved, significant and insignificant at six-months post-examination based on medical record abstraction among participants with indeterminate but potentially clinically significant ECFs (E3/E4s) and participants with pulmonary nodules. Estimate the relationship between participant characteristics and clinically significant findings for participants with E3/E4 ECFs and participants with pulmonary nodules.
Estimate Relative Risk | 6 Months
  Estimate the relative risk of confirmed clinically significant findings within six months of receiving CTC among participants with indeterminate but potentially significant ECFs (E3/E4s) and participants with pulmonary nodules, compared with participants with no ECFs (E1s).
Determine Potential Predictors | 6 Months
  Determine potential predictors associated with increased likelihood of receiving follow-up diagnostic imaging, hospitalization, and interventional procedures within six months of receiving CTC among participants with indeterminate but potentially significant ECFs (E3/E4s), including participants with pulmonary nodules.
Estimate Differences in Cost | 6 Months
  Estimate differences in cost associated with common expected follow-up diagnostic imaging, hospitalizations, and interventional procedures within six months of receiving CTC among participants with indeterminate but potentially significant ECFs (E3/E4s) and participants with pulmonary nodules, compared with participants with no ECFs (E1s).

CONTACTS AND LOCATIONS:
Overall Officials: Hanna M. Zafar, MD, MHS, Principal Investigator — University of Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Johnson CD, Chen MH, Toledano AY, Heiken JP, Dachman A, Kuo MD, Menias CO, Siewert B, Cheema JI, Obregon RG, Fidler JL, Zimmerman P, Horton KM, Coakley K, Iyer RB, Hara AK, Halvorsen RA Jr, Casola G, Yee J, Herman BA, Burgart LJ, Limburg PJ. Accuracy of CT colonography for detection of large adenomas and cancers. N Engl J Med. 2008 Sep 18;359(12):1207-17. doi: 10.1056/NEJMoa0800996. PMID 18799557